CLINICAL TRIAL: NCT03438955
Title: A Two-cohort, Single-sequence, Parallel, Open Label, Multiple Oral Dosing Phase I Study to Evaluate the Safety and the Pharmacokinetic Drug-drug Interaction of Omega-3 and Atorvastatin in Healthy Male Volunteers
Brief Title: Phase I Drug-drug Interaction of Omega-3 and Atorvastatin
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: DongKoo Bio & Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 17OA-15003
Record Dates: First submitted 2018-02-08; First posted 2018-02-20 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Hyperlipidemia, Hypertriglyceridemia
MeSH Terms: conditions — Hyperlipidemias; Hypertriglyceridemia | interventions — Omacor; Telmisartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A (Experimental): Administration of omacor soft capsule 4000mg for 16 days, and followed by omacor soft capsule 4000mg and Pritor tablet 40mg in combination for 7 days.
  Interventions: Drug: Omacor; Drug: Omacor + Pritor
- Cohort B (Experimental): Administration of Pritor tablet 40mg for 7 days, and followed by Pritor tablet 40mg and Omacor soft capsule 4000mg in combination for 16 days.
  Interventions: Drug: Pritor; Drug: Pritor + Omacor

INTERVENTIONS:
Drug: Omacor — Omacor soft capsule 4000mg for 16days
  Arms: Cohort A
Drug: Pritor — Pritor tablet 40mg for 7days
  Arms: Cohort B
Drug: Omacor + Pritor — Omacor soft capsule 4000mg + Pritor tablet 40mg for 7days
  Arms: Cohort A
Drug: Pritor + Omacor — Pritor tablet 40mg + Omacor soft capsule 4000mg for 16dyas
  Arms: Cohort B

SUMMARY:
This study evaluates the safety and pharmacokinetic drug-drug interactions of omega-3 and atorvastatin in healthy male volunteers. Half of the participants will receive omega-3 for 16 days to be steady state of omega-3 and followed by omega-3 and atorvastatin in combination for 7 days. The other half will receive Atorvastatin for 7 days to be steady state of Atorvastatin, and followed by Atorvastatin and Omega-3 in combination for 16 days.

ELIGIBILITY:
Inclusion Criteria:

* 50kg or less of body weight and body mass index of 18 ~ 30kg/m²
* No congenital or chronic disease requiring treatment, and no pathological symptoms or findings as a result of medical examination
* Eligible for the clinical trial as a result of a clinical laboratory test, 12-lead ECG, V/S test at the screening

Exclusion Criteria:

-

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-07-31 (Estimated); Study Completion 2018-08-31 (Estimated)

PRIMARY OUTCOMES:
Cohort A | Day 1 -20hours, -16hours, -12hours, 0hours, Day 13, 14, 15 0hours, Day 16 0, 1, 2, 3, 4, 6, 8, 12, 24hours, Day 23 0, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 14, 24hours
  Area under curve(0-t) of EPA total lipid and Docosahexaenoic acid total lipid AUC t,ss and C max, ss of Atorvastatin
Cohort B | Day 1 0hours, Day 5, 6 0hours, Day 7 0, 0.25 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12 ,24hours, Day 23 0, 0.25, 0.5, 0.75, 1, 1.25, 2, 3, 4, 6, 8, 12, 24hours
  Area under curve(0-t) of Atorvastatin

CONTACTS AND LOCATIONS:
Overall Officials: Min Kyu Park, MD, Principal Investigator — Dong-A National Univ. Hos.
Locations (1):
- Dong-A National University Hospital, Busan, South Korea

IPD SHARING:
Plan to Share IPD: No